CLINICAL TRIAL: NCT01823393
Title: Balloon Aortic Valvuloplasty Performed Without Heparin to Decrease Vascular and Bleeding Complications of the Procedure
Acronym: HEPAVALV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty of inclusion
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9026
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Aortic Stenosis, Non-rheumatic
Keywords: balloon aortic valvuloplasty indication; heparin; hemorrhagic; ischemic
MeSH Terms: conditions — Aortic Valve Stenosis; Ischemia | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heparin (Experimental): injection of unfractionated heparin (50 IU / kg)
  Interventions: Drug: Heparin
- NaCl (Placebo Comparator): without heparin
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Heparin — Valvuloplasty is performed in a conventional manner, ie with an injection of unfractionated heparin (50 IU / kg) at the start of procedure
  Other Names: Unfractioned heparin
  Arms: Heparin
Drug: NaCl — valvuloplasty is performed without heparin (placebo injection)
  Other Names: placebo
  Arms: NaCl

SUMMARY:
To assess if the non use of heparin sodium during balloon aortic valvuloplasty reduces serious complications due to the procedure, by decreasing the rate of vascular and hemorrhagic complications without increasing the rate of ischeamic events.

ELIGIBILITY:
Inclusion Criteria:

* be over 18
* carry a tight and symptomatic aortic stenosis
* have an indication for a ballon aortic valvuloplasty
* Subject have signed his written informed consent

Exclusion Criteria:

* Have an absence of femoral surgical approach
* have a criticial hemodynamic state, considered as outdrove for the treatment
* have a severe aortic failure
* allergia to heparin
* contraindication to heparin or/and local anaesthetic
* be treted by low molecular weight heparin in less than 12 hoursbefore the intervention or by standard heparin in less than 4 hours before the valvulopasty
* have a tight but not symptomatic aortic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2016-10-22 (Actual); Study Completion 2016-10-22 (Actual)

PRIMARY OUTCOMES:
Number of serious complication : vascular, hemorrhagic or ischaemic complication | Up to10 days after the valvuloplasty (D1-D10 after the intervention)

SECONDARY OUTCOMES:
Number of any non serious complication directly associated with the procedure (vascular, hemorrhagic or ischaemic complication) | up to30 days after the valvuloplasty (until D30 after intervention)
  Non serious complication is complication directly associated with the valvuloplasty which could be vascular complications medically treated (compression), BARC 2 hemorrhage, general procedure complications
number of a serious complication : vascular, hemorrhagic or ischaemic complication | up to 30 days after valvuloplasty

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PU PH, Principal Investigator — UH Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France